CLINICAL TRIAL: NCT03163420
Title: Effect of Pre-operative Diclofenac Potassium on the Anesthetic Efficacy of Inferior Alveolar Nerve Block in Cases With Symptomatic Irreversible Pulpitis: A Randomized Controlled Trial
Brief Title: Diclofenac Potassium on IANB Efficacy in Symptomatic Irreversible Pulpitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Ahmed Youssef, Postgraduate student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CEBC-CU-2016-10-149
Record Dates: First submitted 2017-05-15; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2016-10

CONDITIONS: Irreversible Pulpitis
Keywords: Anesthetic efficacy; Diclofenac; Irreversible pulpitis
MeSH Terms: interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): placebo
  Interventions: Other: Placebo
- Diclofenac potassium (Experimental): Diclofenac potassium 50 mg
  Interventions: Drug: Diclofenac potassium

INTERVENTIONS:
Drug: Diclofenac potassium — Diclofenac potassium 50 mg granules for oral solution
  Other Names: Catafast-Novartis International AG, Basel, Switzerland
  Arms: Diclofenac potassium
Other: Placebo — Fructose
  Arms: Placebo

SUMMARY:
The aim of this clinical trial is to evaluate the effect of pre-operative administration of diclofenac potassium on the efficacy of inferior alveolar nerve block on using 2% mepivacaine anaesthetic agent in patients with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
Objective: The aim of this clinical trial is to evaluate the effect of pre-operative administration of diclofenac potassium on the efficacy of inferior alveolar nerve block on using 2% mepivacaine anaesthetic agent in patients with symptomatic irreversible pulpitis.

Design: Randomized double-blind controlled trial.

Setting and conduct:

* Patients source: Out patients of the clinic of Endodontics at the Faculty of Oral and Dental Medicine, Cairo University.
* Patients will be clinically and radiographically examined and their eligibility will be assessed and preoperative pain will be measured. Eligible patients will be treated in one visit.
* Patients will be randomly assigned to one of 2 groups: experimental group (taking a 50 mg diclofenac potassium packet) and the control group (taking a placebo packet). Each packet will be taken 30 minutes before starting treatment. The patient's pain will be assessed before local anesthetic administration using Heft- Parker Visual Analog Scale (HP- VAS). . After 15 minutes of the initial inferior alveolar nerve block (IANB) of 1.8 ml of 2% mepivacaine hydrochloride with 1:100000 epinephrine, the teeth will be examined using a cold pulp sensitivity test; in case of lip numbness together with no or mild pain on cold, the treatment will be initiated.
* During root canal treatment, no to mild pain response on HP- VAS will be considered success. In case of failure, supplemental anesthesia will be administered.
* Main outcome measures: Anesthetic success during root canal treatment using HP VAS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in good health as determined by a medical history and oral questioning. (ASA I or II)
2. Age range is between 18 and 50 years.
3. Patients having symptomatic irreversible pulpitis in one of their mandibular molars.
4. Patients who can understand Heft Parker Visual Analogue Scales VAS.
5. Patients accepting to participate in the study and able to sign informed consent.

Exclusion Criteria:

1. Pregnant female patient.
2. Patients allergic to diclofenac potassium or mepivacaine.
3. Patients having active pain in more than one mandibular molar.
4. Patients who had taken analgesics in the 12 hours preceding the injection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
anesthetic success | Intraoperative
  Pain during treatment is measured using Heft Parker VAS

SECONDARY OUTCOMES:
Pain on injection of initial IANB | Intraoperative
  measured using Heft Parker VAS

CONTACTS AND LOCATIONS:
Overall Officials: Khaled M Ezzat, Professor, Study Director — Faculty of Oral and Dental medicine, Cairo University; Suzan AW Amin, PhD, Study Chair — Faculty of Oral and Dental medicine, Cairo University
Locations (1):
- Faculty of Oral and dental medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prasanna N, Subbarao CV, Gutmann JL. The efficacy of pre-operative oral medication of lornoxicam and diclofenac potassium on the success of inferior alveolar nerve block in patients with irreversible pulpitis: a double-blind, randomised controlled clinical trial. Int Endod J. 2011 Apr;44(4):330-6. doi: 10.1111/j.1365-2591.2010.01833.x. PMID 21692235
- [Background] Shetkar P, Jadhav GR, Mittal P, Surapaneni S, Kalra D, Sakri M, Basavaprabhu A. Comparative evaluation of effect of preoperative alprazolam and diclofenac potassium on the success of inferior alveolar, Vazirani-Akinosi, and Gow-Gates techniques for teeth with irreversible pulpitis: Randomized controlled trial. J Conserv Dent. 2016 Sep-Oct;19(5):390-5. doi: 10.4103/0972-0707.190013. PMID 27656053
- [Background] Saha SG, Jain S, Dubey S, Kala S, Misuriya A, Kataria D. Effect of Oral Premedication on the Efficacy of Inferior Alveolar Nerve Block in Patients with Symptomatic Irreversible Pulpitis: A Prospective, Double-Blind, Randomized Controlled Clinical Trial. J Clin Diagn Res. 2016 Feb;10(2):ZC25-9. doi: 10.7860/JCDR/2016/16873.7195. Epub 2016 Feb 1. PMID 27042580